CLINICAL TRIAL: NCT00213031
Title: A Randomized, Placebo-controlled, Double-blind Trial to Assess Expanded Safety, Acceptability and Preliminary Effectiveness of PC-515 (Lambda Carrageenan) for Vaginal Use as a Possible Microbicide
Brief Title: Safety, Acceptability and Preliminary Effectiveness of PC-515 for Vaginal Use as a Possible Microbicide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Nat'l Cntr. for HIV, STD, & TB Prevention Atlanta: Division of STD Prevention,Div. of HIV/AIDS Prevention-Surveillance & Epidemiology (Unknown); National Center for Infectious Diseases (Other Government); Ministry of Health, Thailand (Other Government); Collaboration (TUC) (Unknown); Chiang Rai Public Health Office (Other Government); Chiang Rai District Health Office (Other Government); Chiang Rai Municipal Health Office (Other Government); Chiang Rai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Population Council #271; CDC & Prevention #2485
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections; Chlamydia Trachomatis; Neisseria Gonorrhoeae; Trichomonas Vaginitis; Syphilis; Herpes Simplex
Keywords: microbicides; HIV prevention; sexually transmitted infections; female-initiated protection; carrageenan; expanded safety trial; HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Trichomonas Vaginitis; Syphilis; Herpes Simplex; Sexually Transmitted Diseases

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
The primary aims of the study were to assess the safety and acceptability of PC-515 when applied vaginally at least three times weekly for 12 months. Secondary aims were to gather preliminary data on Carraguard's effectiveness in preventing male-to-female transmission of HIV, and other STIs.

The hypothesis was that Carraguard would cause little or no significant irritation, including lesions; and that women would find Carraguard acceptable. The study was not powered to determine effectiveness, but based on safety, acceptability and feasibility parameters, the outcome of the Phase 2 trial would enable a decision whether or not to proceed to a Phase 3 trial.

DETAILED DESCRIPTION:
Carraguard™ (PC-515), the Population Council's lead candidate microbicide, was tested in a triple-masked, randomized, placebo-controlled trial fielded in one site in Chiang Rai, northern Thailand. The primary aims of the study were to assess Carraguard's safety (toxicity) - including signs of local irritation, such as itching or burning; changes in vaginal flora; and incidence of abnormal external genital, vaginal, and cervical findings - when applied vaginally for 12 months; to evaluate acceptability; to assess feasibility of conducting a large scale microbicide trial in a non-sex worker population; to gauge women's reactions to a non-contraceptive microbicide; and to explore microbicide use dynamics in a Thai population.

Secondary aims were to investigate HIV infections averted (preliminary indications); other sexually transmitted infections averted - including C. trachomatis, N. gonorrhoeae, T. vaginalis, and T. pallidum (preliminary indications); and effect on cervical cytology.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by medical history, physical examination and results of laboratory screening tests
* Aged 18 years or older
* Resident in the area for at least one year and planning to stay for at least 12 months
* HIV-seronegative at baseline
* Willing and able to comply with the study protocol (including being tested for HIV, learning the results, and undergoing clinical evaluations)
* Able to achieve a score of 80% or better on true-false test of key study concepts
* Able to give informed consent

Exclusion Criteria:

* Pregnant or desire to become pregnant at time of study participation
* Delivered or aborted a pregnancy within the six weeks prior to screening
* Male sex partner known at enrollment to be HIV positive
* History of surgery on external genitalia, vagina or cervix in the six weeks prior to screening
* Recent history of non-menstrual vaginal bleeding with intercourse
* Clinically detectable genital abnormality (including presence of warts, or a structural or congenital abnormality)
* Clinical suspicion of a reproductive tract infection (RTI), defined as the presence of a genital ulcer visible to the naked eye, an abnormal vaginal discharge or purulent cervicitis, or untreated positive STD result (Women could be enrolled after treatment of identified RTI. Women with persistent genital epithelial disruption, i.e., ulcer, abrasion or fissure, were not eligible.
* Women with other persistent abnormal signs, such as vaginal or cervical discharge, despite treatment of identified RTI, were eligible)
* Abnormal Pap smear (Class II or above)
* History of sensitivity/allergy to latex
* Concurrent participation in another trial of a vaginal product
* Injection of recreational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2000-02 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Safety: Genital exam & interview for symptoms after 14 days & monthly thereafter; colposcopy done throughout trial at clinicians' discretion; monthly testing to detect changes in vagina flora.
Compliance: collection of applicators and interview(monthly)
Acceptability: interview (quarterly)

SECONDARY OUTCOMES:
Preliminary effectiveness: Swabs taken to test for sexually transmitted infections - gonorrhea, chlamydia, trichomoniasis and for genital ulcer disease, if ulceration was detected; blood drawn for syphilis and HIV testing and for HSV-2 Pap smear to det

CONTACTS AND LOCATIONS:
Overall Officials: Janneke HMM van de Wijgert, Ph.D., Principal Investigator — Population Council
Locations (1):
- Chiang Rai Health Club, Chiang Rai, Thailand